CLINICAL TRIAL: NCT06452706
Title: The Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQB2102 for Injection in Human Epidermal Growth Factor Receptor 2 (HER2) Negative Recurrent/Metastatic Breast Cancer
Brief Title: The Clinical Trial of TQB2102 for Injection Against Human Epidermal Growth Factor Receptor 2 Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-II-02
Record Dates: First submitted 2024-06-06; First posted 2024-06-11 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2102 for injection (Experimental): 7.5mg/kg TQB2102, intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle.
  Interventions: Drug: TQB2102 for injection

INTERVENTIONS:
Drug: TQB2102 for injection — TQB2102 for injection is a HER2 dual-antibody-drug conjugate (ADC).

SUMMARY:
This study aims to evaluate the efficacy and safety of TQB2102 for injection in HER2 negative recurrent/metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* The participants voluntarily participate in the study and sign an informed consent form.
* Age: 18-75 years old; Eastern Cooperative Oncology Group (ECOG) score: ≤1 point; Expected survival period exceeds 3 months.
* Breast cancer patients diagnosed as HER2 negative by pathology, with evidence of local recurrence or distant metastasis are not suitable for surgery or radiation therapy aimed at healing.
* Sufficient tumor tissue samples must be available for HER2 evaluation by pathologists at the main research center.
* The participants's previous treatment needs to meet the following criteria: failure after receiving at least first-line systemic chemotherapy during the recurrence /metastasis stage (for hormone receptor positive participants, failure after receiving cyclin-dependent kinase 4 and 6 (CDK4/6) inhibitors combined with endocrine therapy during the recurrence/metastasis stage.
* There exists disease progression or intolerance during or after the most recent treatment before enrollment.
* According to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 standard, there should be at least one measurable lesion.
* The main organ functions well and meets certain standards.
* Female participants of childbearing age should agree to use contraceptive measures during the study period and within 6 months after the end of the study; within 7 days prior to enrollment, the serum pregnancy test was negative and must be a non lactating subject; male participants should agree to adopt avoidance measures during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* Concomitant diseases and medical history:

  1. Have experienced or currently suffer from other malignant tumors within 5 years prior to the first medication use;
  2. Uncontrollable toxic reactions above CTCAE level 1 caused by any previous treatment;
  3. Received significant surgical treatment or significant traumatic injury within 28 days prior to the first medication use;
  4. Long term unhealed wounds or fractures;
  5. Participants who have a history of interstitial lung disease/pneumonia (non infectious) requiring steroid intervention treatment in the past, or currently have interstitial lung disease/pneumonia, or whose screening imaging suggests suspected interstitial lung disease/pneumonia and cannot be ruled out;
  6. An arterial/venous thrombotic event occurred within 6 months prior to the first medication use;
  7. Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders;
  8. Subjects with any severe and/or uncontrolled diseases. Rheumatoid arthritis with joint function activity graded as Grade IV or requiring wheelchair or bed rest.
* Tumor related symptoms and treatment:

  1. Participants who have received other anti-tumor drug treatments such as chemotherapy, curative radiotherapy, or immunotherapy within 4 weeks before the first medication, or who are still within the 5 half-lives of the drug (whichever is the shortest); Participants who have previously received local radiotherapy;
  2. Received endocrine therapy or traditional Chinese patent medicines and simple preparations with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug directions within 2 weeks before the first drug use;
  3. Imaging shows that the tumor has invaded important blood vessels, or the researcher determines that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies;
  4. Uncontrollable pleural effusion, ascites, and moderate or higher amounts of pericardial effusion that require repeated drainage;
  5. Known presence of cancerous meningitis or clinically active central nervous system metastasis;
  6. Severe bone damage caused by tumor bone metastasis. Suffering from lung diseases that have been determined by the researcher to be unsuitable for participation in this study.
* Individuals who are known to be allergic to the investigational drug or its excipients, or allergic to humanized monoclonal antibody products.
* Individuals who have participated in and used other anti-tumor clinical trial drugs within 4 weeks prior to the first medication use.
* According to the judgment of the researchers, there are situations that seriously endanger the safety of the subjects or affect their completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 24 months after study start.
  The percentage of subjects achieving complete response (CR) or partial response (PR) as assessed by the investigator based on the RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival | Up to 36 months after study start
  From randomization to the time of disease progression or death, whichever occurs first.
Duration of disease remission | Up to 24 months after study start
  For subjects whose best response is CR or PR , it is defined as from the date when tumor response is first recorded to the date when disease progression is first recorded or the date of death from any cause, whichever occurs first.
Disease control rate | Up to 24 months after study start
  Percentage of subjects with CR, PR, or stable disease(SD) at 6 weeks or more as determined by RECIST 1.1.
Clinical benefit rate | Up to 24 months after study start
  The percentage of subjects achieving CR, PR or SD as assessed by the investigator based on the RECIST 1.1.
Overall survival | Up to 48 months after study start
  From randomization to the time of death from any cause.
Incidence of adverse events | Up to 36 months after study start
  All adverse medical events (e.g. adverse events, serious adverse event and abnormal laboratory values) that occurred after the subject received the investigational drug.
Anti-drug antibody (ADA) | 1 hour Before infusion on Cycle 1 Day1, Cycle 2 Day1, Cycle 4 Day1, Cycle 7 Day1, Cycle 12 Day1, and 30 days after the end of the last infusion. Each cycle is 21 days
  Incidence of ADA
HER2 | Up to 24 months after study start
  Correlation analysis between HER2 expression level and TQB2102 treatment response
circulating tumor DNA (ctDNA) | Up to 24 months after study start
  Exploring the genetic variation and dynamic changes of ctDNA, including ctDNA clearance。

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Bozhou People's Hospital, Bozhou, Anhui
  - Chuzhou First People's Hospital, Chuzhou, Anhui
  - Anhui Provincial Public Health Clinical Center, Hefei, Anhui
  - Ma'anshan People's Hospital, Ma’anshan, Anhui
  - Wuhu Hospital Affiliated to East China Normal University, Wuhu, Anhui
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The Third People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The First People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - Ruijin Hospital ,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Cancer Hospital Affiliated to Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Suzhou Municipal Hospital, Suzhou, Zhejiang
  - Wenzhou Medical University Affiliated First Hospital, Wenzhou, Zhejiang